CLINICAL TRIAL: NCT05369026
Title: Effect of Fortetropin Supplementation in Young Men During Muscle Disuse
Brief Title: Effect of a Natural Source Supplementation on Muscle Mass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Myos Corporation (Unknown)
Responsible Party: Principal Investigator, Stuart Phillips, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 7935
Record Dates: First submitted 2022-05-03; First posted 2022-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Muscle Disuse Atrophy; Nutrition, Healthy
Keywords: Skeletal muscle; Supplementation; Disuse; Single-leg immobilization
MeSH Terms: conditions — Muscular Disorders, Atrophic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fortetropin (Experimental): Foretetropin, which is non-thermal pasteurized, freeze-dried fertilized egg yolk, per day
  Interventions: Other: Single leg immobilization
- Placebo (Placebo Comparator): Cheese powder, which is isonitrogenous, isoenergetic, and macronutrient-matched with Fortetropin
  Interventions: Other: Single leg immobilization

INTERVENTIONS:
Other: Single leg immobilization — 2 weeks of single-leg immobilization

SUMMARY:
Periods of muscle disuse are commonly experienced in young and elderly individuals as a result of short-term hospitalization or leg casting after injury. Periods of immobilization result in a profound loss of muscle mass and strength. This loss of muscle mass can have negative effects on health and the ability to carry out activities of daily living. Thus, it is very important to try to maintain muscle mass during muscle disuse. Recent research suggests that Fortetropin, which is an all-natural protein-fat complex made from fertilized hen egg yolks, can enhance muscle mass and strength with weightlifting in young men. In this study, we aim to investigate the safety and tolerability of Fortetropin and whether Fortetropin supplementation can reduce or prevent the loss of muscle mass during single-leg immobilization while you are wearing a knee brace. To make this decision, we require a study to compare Fortetropin to a placebo (something that contains the same amount of protein and energy as Fortetropin). The findings from this study will help us understand if Fortetropin supplementation is safe, tolerable, and can be used to slow muscle loss in people who undergo periods of muscle disuse (i.e. surgery, sickness).

ELIGIBILITY:
Inclusion Criteria:

* Men, between the ages of 20-25 years (inclusive).
* Willing and able to provide informed consent.
* Be in general good health, non-smoking.
* Body mass index (BMI) between 20-35kg/m2.
* Agree to not consume eggs for the duration of the study.

Exclusion Criteria:

* Use of tobacco related products.
* Veganism or vegetarianism.
* Subject has any concurrent medical, orthopedic, or psychiatric condition that, in the opinion of the investigator, would compromise his/her ability to comply with the study requirements.
* History of cancer within the last 5 years, except basal cell carcinoma, non-squamous skin carcinoma, prostate cancer or carcinoma in situ with no significant progression over the past 2 years.
* Significant orthopedic, cardiovascular, pulmonary, renal, liver, infectious disease, immune disorder (requiring ongoing medical care), or metabolic/endocrine disorder (e.g. diabetes, high cholesterol, elevated fasting blood sugar) or other disease that would preclude oral protein supplement ingestion and/or assessment of safety and study objectives.
* Any cachexia-related condition (e.g. relating to cancer, tuberculosis or human immunodeficiency virus infection and acquired immune deficiency syndrome) or any genetic muscle diseases or disorders.
* Current illness with could interfere with the study (e.g. prolonged severe diarrhea, regurgitation, difficulty swallowing).
* Subject participated in a study of an investigational product less than 60 days or 5 half-lives of the investigational product, whichever is longer, before enrollment in this study.
* Hypersensitivity to any of the components of the test product.
* Excessive alcohol consumption (>21 standard drinks/week, e.g. 18oz glass of 5% beer - 1.5 standard drinks, a 750ml bottle of 12% wine = 5 standard drinks).
* Known sensitivity or allergy to amino acids or any ingredient in the test formulations. 12) Prior gastrointestinal bypass surgery (Lapband, etc.), irritable bowel disease or irritable bowel syndrome.
* History of bleeding diathesis, platelet or coagulation disorders, or antiplatelet/anti-coagulation therapy (up to 81 mg of baby aspirin per day taken as a prophylactic is permitted).
* Personal or family history of clotting disorder or deep vein thrombosis. Deep vein thrombosis is a serious, and potentially lethal, medical condition, therefore, it is imperative if you have personal or family history it is disclosed this to the research staff.
* Concomitant use of corticosteroids, testosterone replacement therapy (ingestion, injection, or transdermal), any anabolic steroid, creatine, whey protein supplements, casein or branched-chain amino acids (BCAAs) within 45 days prior to screening.

Ages: 20 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
Vastus lateralis cross sectional area | Baseline (Day 0), pre-immobilization (Day 14), post-immobilization (Day 28), post-recovery (Day 42)
  Changes in vastus lateralis cross sectional area (CSA) by ultrasonography.
Single fiber cross sectional area | Baseline (Day 0), pre-immobilization (Day 14), post-immobilization (Day 28), post-recovery (Day 42)
  Fiber type dependent single fiber CSA analyzed by immunohistochemistry
Fat-and-bone free-mass | Baseline (Day 0), pre-immobilization (Day 14), post-immobilization (Day 28), post-recovery (Day 42)
  Fat-and-bone free-mass using DXA.

SECONDARY OUTCOMES:
Myostatin level in plasma | Baseline (Day 0) and Post-recovery (Day 42)
  Changes in Myostatin circulation level in plasma.
Leg strength | Baseline (Day 0), pre-immobilization (Day 14), post-immobilization (Day 28), post-recovery (Day 42)
  Changes in isometric muscle strength using Biodex
Basic metabolic panel and liver enzyme | Baseline (Day 0), post-recovery (Day 42)
  Changes in Basic metabolic panel and liver enzyme (ALT and AST) in plasma
Myostatin positive satellite cells | Baseline (Day 0), pre-immobilization (Day 14), post-immobilization (Day 28), post-recovery (Day 42)
  Changes in the number of myostatin positive satellite cells.
Gastrointestinal response to ingestion of the supplement | Pre-immobilization (Day 14), post-immobilization (Day 28), post-recovery (Day 42)
  Assessment of gastrointestinal response to ingestion of the supplement using Likert scale questionnaire. The minimum (best) value is 1 and maximum (worst) value is 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise Metabolism Research Laboratory, McMaster Univeristy, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lim C, McKendry J, Giacomin T, Mcleod JC, Ng SY, Currier BS, Coletta G, Phillips SM. Fortetropin supplementation prevents the rise in circulating myostatin but not disuse-induced muscle atrophy in young men with limb immobilization: A randomized controlled trial. PLoS One. 2023 May 23;18(5):e0286222. doi: 10.1371/journal.pone.0286222. eCollection 2023. PMID 37220119